CLINICAL TRIAL: NCT02465619
Title: To Study and Compare the Clinical Course and Development of Organ Failure in Severe Acute Hepatitis Without Ascites, Non-cirrhotic and Cirrhotic Patients With Ascites [Acute on Chronic Liver Failure] and Acute Deterioration of Previously Decompensated Cirrhosis.
Status: Withdrawn | Type: Observational
Why Stopped: Due to lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-002
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-01

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Severe acute hepatitis: Severe acute hepatitis without ascites.
- Non-cirrhotic
- Cirrhotic patients with ascites
- decompensated cirrhosis

SUMMARY:
The study will be conducted on patients admitted to Department of Hepatology from MARCH 2015 to DECEMBER 2016 at ILBS, New Delhi.All patients presenting to ILBS fulfilling the inclusion criteria will be included in the study and will be categorized and evaluated. The patient will followed over a period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients presenting to hospital with bilirubin ≥5 and INR≥1.5
* Cirrhosis with or without Decompensation presenting with acute deterioration in less than 3 month

Exclusion Criteria:

* Cirrhosis with chronic decompensation.
* Patient on anticoagulant
* Hepatocellular carcinoma
* Septic shock
* Post-liver transplant or resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Cirrhosis: based on previous liver biopsy if available or based on clinical, imaging.
  2. Severe acute hepatitis [14]: fulfilling any 2 of the 3 criteria:
     * Hepatic encephalopathy,
     * Serum bilirubin equal to or more than 10 mg/dl
     * International normalized ratio (INR) more than or equal to 1.6
  3. Acute on chronic liver failure [3]: Acute hepatic insult manifesting as jaundice (serum bilirubin ≥ 5mg/dL) and coagulopathy (INR ≥ 1.5), complicated within 4 weeks by ascites and/or encephalopathy in patients with previously diagnosed or undiagnosed chronic liver disease/cirrhosis, and is associated with a high 28-day mortality.
  4. Acute deterioration of decompensated cirrhosis [4]: Acute decompensation of cirrhosis in the form of one or more major complications of liver disease, including ascites, hepatic encephalopathy, gastrointestinal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Survival | 28 days

SECONDARY OUTCOMES:
Survival | 3 months
total number of patients underwent Transplantation | 3 months
Mortality | 3 months
Number of patients develop liver failure. | 3 months
Number of patients develop SIRS (Systemic Inflammatory Response Syndrome). | 3 months
Number of patients develop sepsis. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India